CLINICAL TRIAL: NCT04266431
Title: EMPOWER Men to Reduce Weight and Inhibit Prostate Cancer Progression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: American Cancer Society, Inc. (Other); Maryland Cigarette Restitution Fund (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: J1976; Rsg-18-147-01-Cce (Other Grant/Funding Number: American Cancer Society); IRB00221103 (Other: Johns Hopkins School of Medicine IRB)
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible consented men will be stratified for randomization according to prostate specific antigen doubling time (PSADT; <6 months or 6-12 months) calculated using 3 values (≥1 week apart; ≤ 3 months from randomization; Memorial Sloan Kettering Cancer Center prediction tool: http://nomograms.mskcc.org/Prostate/PsaDoublingTime.aspx), and body mass index (BMI) at baseline (25 kg/m2 ≤BMI <30 kg/m2 or BMI≥ 30 kg/m2). Following stratification, men will be randomized 1:1 using a computer-generated, password protected randomization enrollment system by the biostatistician. Men will be informed of the random assignment after consenting to the study and completing the baseline questionnaires and blood collection. Study visits will take place at 6 months, 12 months, and 24 months after baseline.
Who Masked: Outcomes Assessor
Masking Description: The randomization scheme will be generated by the senior biostatistician, and access will be restricted for the duration of the trial. The participants and interventionists will not be blinded to study arm. The study staff involved in data collection, staff involved in laboratory measurements, and the biostatistician conducting the data analysis will be blinded to the random assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMPOWER (Experimental): EMPOWER is a multichannel, behavioral lifestyle intervention delivered remotely. The goals of EMPOWER are to induce a loss of 5% or more of initial weight within 6 months and to maintain these improvements at 12 and 24 months, by meeting dietary and physical activity goals. Coach-participant contacts will occur by phone and email, without in-person visits. Coaching contacts will be weekly for the first 12 weeks and then monthly thereafter. Men will have access to a web-based system that (1) provides support for behavioral methods of weight management and (2) allows coaches to review participant self-monitoring data and monitor participant progress towards goals. Men will record diet, exercise, and weight on the web or on a smart phone application.
  Interventions: Behavioral: EMPOWER
- Standard of Care (No Intervention): Men randomized to the standard of care group will continue to receive treatment from the mens' medical oncologist. These men will also be provided with a one page informative brochure on lifestyle recommendations adapted from the American Cancer Society Prostate Cancer Survivorship Care Guidelines, at the time of randomization. At the end of the trial, men in this arm will be offered a one-time counseling session with an intervention coach on healthy lifestyle.

INTERVENTIONS:
Behavioral: EMPOWER — Behavioral weight loss intervention
  Arms: EMPOWER

SUMMARY:
This study will evaluate whether a lifestyle intervention focused on weight loss, EMPOWER, reduces prostate cancer progression at 12 months among men with biochemical recurrence following local treatment for prostate cancer. Half of the men will be randomized to receive the EMPOWER intervention, while the other half will receive standard of care.

DETAILED DESCRIPTION:
Approximately 500,000 US men are living with biochemical recurrent prostate cancer (BCR). Therapies are needed to delay the appearance of metastatic disease and need for androgen deprivation therapy (ADT), which has significant adverse side effects. Observational evidence suggests that weight loss may slow the rate of disease progression. The EMPOWER trial will use an enhanced version of a remote weight loss intervention shown to yield clinically significant weight loss to test whether weight loss reduces prostate cancer progression at 12 months. EMPOWER has the potential to provide men with BCR a "first line therapy" to slow disease progression and delay the need for ADT. Importantly, this "treatment" is without significant side effects, and can improve overall health.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign consent form
* Able to adhere to study protocol
* Demonstrated use of internet and email
* Access to internet at least 4 days per week
* Willingness to change diet, physical activity and weight
* Willingness to be randomized to immediate start or standard of care
* Histologically confirmed diagnosis of adenocarcinoma of the prostate with evidence of biochemical recurrence following local therapy (surgery and radiation will be allowed). Biochemical recurrence will be defined as a PSA >= 0.2 ng/mL.
* Surgically treated men must not be eligible for or decline salvage radiation. Men who recurred within 3 years of completion of salvage radiation will be included.
* Definitive therapy (surgery or radiation) should be at least 4 weeks from time of consent.
* Men who received prior hormone therapy with definitive local therapy (standard with radiation) are permitted if serum testosterone level is >150 ng/dL and hormone treatment was discontinued > 1 year from time of enrollment.
* Body mass index >= 25 kg/m2
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Willingness to return for clinical visit at 6 months, 12 months, and 24 months
* Men receiving testosterone replacement therapy will be included if they are on a stable dose with testosterone levels in the normal range.

Exclusion Criteria:

* Any clinical or radiographic evidence of metastatic disease by computed tomography (CT) of the chest, abdomen and pelvis and technetium-99 bone scintigraphy (bone scan)
* MI, stroke or ASCVD procedure within 6 months
* Serious medical condition likely to hinder accurate measurement of weight, or for which weight loss is contraindicated, or which would cause weight loss
* Unstable angina or medical conditional that would prevent routine exercise
* Prior or planned bariatric surgery
* Use of prescription weight loss medication (including off label use of medications) or over-the-counter orlistat within 6 months
* Chronic use (at least past 6 months) of medications likely to cause weight gain or prevent weight loss (e.g. corticosteroids, lithium, olanzapine, risperidone, clozapine), including androgen deprivation therapy
* Unintentional or intentional weight loss within 6 months of enrollment (≥ 5% of body weight)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Proportion of men who develop prostate specific antigen (PSA) progression or radiographic progression | 12 months
  Proportion of men who develop prostate specific antigen (PSA) progression or radiographic progression (e.g. soft tissue or bone lesions). In accordance with the Prostate Cancer Clinical Trials Working Group (PCWG2) criteria, PSA progression will be defined as an increase that is ≥25% and ≥2 ng/mL above the nadir that is confirmed by a second value in ≥3 weeks, soft tissue lesions will be defined using RECIST 1.1 criteria, and bone lesions will be defined as ≥2 new lesions, with a confirmatory scan ≥6 weeks later.

SECONDARY OUTCOMES:
Proportion of men who experience clinical progression | Up to 24 months
  Proportion of men who experience clinical progression defined as development of (1) pain that, in the medical oncologist's opinion, is secondary to prostate cancer, or (2) a pathologic fracture or other skeletal event.
PSA doubling time | Up to 24 months
  PSA doubling time calculated using 3 values (≥1 week apart; Memorial Sloan Kettering Cancer Center prediction tool)
Change in PSA | 6 months, 12 months, and 24 months
  Change in PSA level (ng/mL).

OTHER OUTCOMES:
Change in weight | 6 months, 12 months, and 24 months
  Weight measured by scale in kilograms (kg).
Change in waist circumference | 6 months, 12 months, and 24 months
  Waist circumference [in centimeters (cm)] using an anthropometric measuring tape at a horizontal plane that is one cm above the navel.
Change in diet | 6 months, 12 months, and 24 months
  Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24)
Change in physical activity | 6 months, 12 months, and 24 months
  Community Healthy Activities Model Program for Seniors (CHAMPS) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Joshu, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 6 months after publication
Access Criteria: Investigators interested in using study data to address questions beyond the scope of the project can request de-identified data from the PI in writing. The PI will provide access to de-identified data if the study goals are consistent with participant consent, and the requesting investigative team can provide the necessary assurances of proper handling of the data, including Institutional Review Board (IRB) approval and execution of a data use agreement.